CLINICAL TRIAL: NCT07127029
Title: Effect Of Petrolatum On Absorption of Fast Gut Suture In Vivo
Brief Title: Effect of Petrolatum Coating on Fast-absorbing Gut Suture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Antonio Uniformed Services Health Education Consortium (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jason Susong, Principal Investigator, San Antonio Uniformed Services Health Education Consortium
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: FWH20160040H
Record Dates: First submitted 2025-08-08; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Suture; Suture Dermatologic; Mohs Micrographic Surgery; Suture Techniques; Dermatology; Closure Technique; Absorbable, Coated Sutures
Keywords: Petrolatum; Absorbable Suture; Gut Suture; Fast-absorbing Gut Suture; Wound Closure; Suture Coating

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 6-0 Fast-Absorbing Gut Suture (Experimental): Two 6-0 fast-absorbing gut sutures were placed in the skin of deltoid, randomized to site A/B for the control (uncoated) and intervention (petrolatum coated) suture.
  Interventions: Device: Petrolatum coating of fast-absorbing gut suture

INTERVENTIONS:
Device: Petrolatum coating of fast-absorbing gut suture — 6-0 fast absorbing gut suture was coated with sterile petrolatum and a single interrupted suture was placed into the skin of the deltoid
  Other Names: petrolatum coating

SUMMARY:
This study is designed to evaluate the effect of using petrolatum to coat gut suture. This coating is commonly performed to make the suture more easy to handle; however, it was unknown if it affects the absorption rate of the suture. Two gut sutures were placed into the skin of 14 healthy volunteers and randomized between coated and uncoated with petrolatum. Participants self-reported the time to resorption. The study concluded that there was no significant effect to the application of petrolatum, and reinforced that the gut sutures are a natural product with some inherent variability to their absorption.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers within department of Dermatology
* Able to receive care within the host facility (Dept of Defense)

Exclusion Criteria:

* current or planned pregnancy
* Allergy to lidocaine
* Infection on the shoulder site

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2016-10-14 (Actual); Study Completion 2016-10-14 (Actual)

PRIMARY OUTCOMES:
Length of time that suture remains intact in skin following petrolatum coating compared with standard fast-absorbing gut suture. | Postprocedurally daily until suture is degraded (less than 2 weeks)
  Length of time in hours of suture remaining in skin prior to breakdown was recorded for both uncoated and coated suture.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Susong JR, Neiner JR. Effect of petrolatum coating on fast-absorbing gut suture. J Am Acad Dermatol. 2018 Nov;79(5):952-953. doi: 10.1016/j.jaad.2018.04.041. Epub 2018 Apr 30. No abstract available. PMID 29723559